CLINICAL TRIAL: NCT05386823
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study Following Intravenous Administration of HF1K16 in Healthy Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of HF1K16
Brief Title: Evaluate the Safety, Tolerability and PK of HF1K16 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HighField Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HF1K16-101
Record Dates: First submitted 2022-03-16; First posted 2022-05-23 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 3 mg/m² HF1K16 (Experimental)
  Interventions: Drug: HF1K16
- 6 mg/m² HF1K16 (Experimental)
  Interventions: Drug: HF1K16
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HF1K16 — HF1K16 for Injection doses will be calculated based on subject weight measured at admission, and diluted in sterile saline (0.9% sodium chloride). Doses will be administered using an IV infusion pump over a period of approximately 60 minutes at 2.5 mL/min.
  Arms: 3 mg/m² HF1K16; 6 mg/m² HF1K16
Drug: Placebo — Placebo will be sterile saline (0.9% sodium chloride) which will be administered using an IV infusion pump over a period of approximately 60 minutes at 2.5 mL/min.
  Arms: Placebo

SUMMARY:
HF1K16 is an investigational pegylated liposome formulation of tretinoin for injection for the treatment of solid tumors through targeting myeloid derived suppressor cells (MDSCs). This phase 1 Trial is a Randomized, Double-Blind, Placebo-Controlled Study in Healthy Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of HF1K16.

DETAILED DESCRIPTION:
Tretinoin is a naturally occurring vitamin A metabolite that participates in many biological processes. It is not a cytolytic agent but instead induces cytodifferentiation and decreased proliferation of APL cells achieving complete remission (CR). In addition, ATRA and similar retinoids were also discovered to have significant immune-modulating activities towards Myeloid derived suppressor cells (MDSCs) that contribute greatly to cancer growth and progression. Preclinical efficacies of HF1K16 to induce MDSC differentiation into dendritic cells (DCs) and downregulate their inhibitory effects on cytotoxic T cell activities against cancer have been demonstrated.

HF1K16 is a pegylated liposome formulation of tretinoin developed for improved PK behavior, higher therapeutic index, and more specific targeted mechanism towards MDSCs. The objectives of this study are to assess the safety and tolerability of HF1K16. The ATRA pharmacokinetic parameters will be determined with correlations to the liposome doses administered.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent and complying with study procedures;
2. Between the ages of 18 and 55 years, inclusive;
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive and body weight not less than 50 kg;
4. Female subjects must have a negative pregnancy test result at screening and at admission;
5. Female subjects are:

   1. Surgically sterile for at least 3 months prior to screening by one of the following means:

      * Bilateral tubal ligation
      * Bilateral salpingectomy (with or without oophorectomy)
      * Surgical hysterectomy
      * Bilateral oophorectomy (with or without hysterectomy)
   2. Postmenopausal, defined as the following:

      * Last menstrual period greater than 12 months prior to screening, and
      * Postmenopausal status confirmed by serum follicle stimulating hormone (FSH) and estradiol levels at screening;
6. Male subjects must agree to utilize a highly effective method of contraception (condom plus spermicide) during heterosexual intercourse from the time of clinic admission until 12 weeks following the end of study visit, and refrain from donating sperm for this same period;
7. Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, 12-lead ECG, and vital signs;
8. Have clinical laboratory renal (eGFR, creatinine) and liver (AST, ALT, Total bilirubin) function within normal range and other clinical laboratory results within normal range or outside normal range assessed as clinically non-significant by the Investigator at screening and admission;
9. Non-smoker and has not been exposed to any products containing nicotine in the last 6 months;
10. Willing and able to adhere to study restrictions and to be confined at the Clinical Research Unit

Exclusion Criteria:

1. Clinically significant reported history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
2. Known or suspected malignancy;
3. Reported history of pancreatitis or gall stones;
4. Reported history of unexplained syncope, symptomatic hypotension or hypoglycemia;
5. Reported family history of long QTc syndrome or a QTc of > 450 ms at screening;
6. Reported history of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance;
7. Poor venous access;
8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV) at screening;
9. Donated or lost >500 mL of blood in the previous 3 months prior to screening;
10. Taken an investigational drug or participated in a clinical trial within 30 days (or 5 half-lives) prior to first dose of study drug, whichever is longer;
11. Taken any prescription medications within 14 days or 5 half-lives (whichever is longer) of the first dose of study drug;
12. Taken any prescription or non-prescription drugs and herbal medication known to be CYP450 inducers, inhibitors, and substrates within 14 days prior to screening (See Appendix B);
13. Taken daily Vitamin A supplement within 3 months prior to screening;
14. Major surgery or hospitalization within 6 months prior to screening that in the Investigators opinion would put the subject or study conduct at risk;
15. A history of prescription drug abuse, or illicit drug use within 9 months prior to screening;
16. A history of alcohol abuse according to medical history (≥ 2 drinks per day for male and ≥ 1 drink per day for female) within 9 months prior to screening;
17. A positive screen for alcohol, drugs of abuse at screening or admission;
18. An unwillingness or inability to comply with food and beverage restrictions during study participation;
19. Use of over-the-counter (OTC) medication within 7 days, and/or herbal medications (including herbal teas, garlic extracts) within 7 days prior to first dose of study drug;
20. Have a history of allergic reactions (either spontaneous or following drug administration) to ATRA or to any of the excipients or related compounds, including vitamin A;
21. Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tracey, MD, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol and SAP
Supporting Information: Study Protocol, SAP
Time Frame: six month after completion
Access Criteria: public

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen subjects were enrolled and randomized to receive active study drug or placebo. All subjects were recruited in medical clinic,Frontage Clinical Services, Inc. started on 20March2021 till 28July2021.
Groups:
- 3 mg/m² HF1K16: 6 subjects received 3 mg/m² of study drug
- 6 mg/m² HF1K16: 6 subjects received 6 mg/m² of study drug
- Placebo: 4 subjects received placebo
Period: Overall Study
Arm/Group | 3 mg/m² HF1K16 | 6 mg/m² HF1K16 | Placebo
Started | 6 | 6 | 4
Completed | 6 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 3 mg/m² HF1K16: 6 subjects received 3 mg/m² of HF1K16
- 6 mg/m² HF1K16: 6 subjects received 6 mg/m² of HF1K16
- Total: Total of all reporting groups
Arm/Group | 3 mg/m² HF1K16 | Placebo | 6 mg/m² HF1K16 | Total
Number analyzed (Participants) | 6 | 4 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 6 | 16
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 6 | 4 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 3 | 4 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 3 | 10
  White | 3 | 0 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
age [Mean (Full Range); unit: years] | 37.3 [30 to 48] | 47.3 [32 to 55] | 40 [26 to 48] | 40.8 [26 to 55]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Event (AE) and Severe Adverse Event (SAE)
Description: Safety evaluation within 8 days after first dose, including frequency of adverse event (AE) and severe adverse event (SAE)
Time Frame: from Day 1 to Day 8
Population: The analysis population included all participants who exposure to study drug
Measure: Number; unit: participants
Groups:
- Placebo: The subjects received single IV doses of placebo on Day 1
- HF1K16-3mg/m²: Cohort 1: The subjects received 3 mg/m² single IV doses of HF1K16 on Day 1
- HF1K16-6mg/m²: Cohort 2: The subjects received 6 mg/m² single IV doses of HF1K16 on Day 1
Arm/Group | Placebo | HF1K16-3mg/m² | HF1K16-6mg/m²
Number analyzed (Participants) | 4 | 6 | 6
participants
  Number of AEs | 0 | 0 | 4
  Subjects with SAE | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT is defined as Specify that any one grade ≥ 3 AE will halt dose escalation unless the AE is clearly and incontrovertibly due to extraneous causes; Specify that any two grade ≥ 2 AEs will halt dose escalation unless the AEs are clearly and incontrovertibly due to extraneous causes；Grade 3 asymptomatic laboratory abnormalities that resolved to ≤ grade 1 within 3 days may be excluded from the definition of DLT
Time Frame: from Day 1 to Day 8
Population: Analysis population includes all participants who received at least one dose of HF1K16 and completed safety follow-up through the DLT evaluation period
Measure: Number; unit: participants
Arm/Group | HF1K16-3mg/m² | HF1K16-6mg/m²
Number analyzed (Participants) | 6 | 6
participants | 0 | 0

3. Secondary Outcome: Peak Drug Concentration (Cmax) After Single Dose of HF1K16
Description: To evaluate pharmacokinetic parameters of free tretinoin and liposome encapsulated tretinoin (4-oxotretinoin) in plasma after single administration of HF1K16
Time Frame: pre-infusion (within 60 minutes prior to the start of infusion) and 0.5, 1, 1.5, 2, 4, 6, 9, 12, 24, 36, and 48 hours relative to start of infusion
Population: The PK analysis population included all participants who were compliant with the study procedures and provided sufficient plasma concentrations of tretinoin and 4-oxotretinoin
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HF1K16-3mg/m² | HF1K16-6mg/m²
Number analyzed (Participants) | 6 | 6
ng/mL
  Cmax of tretinoin | 198 (45.6) | 409 (52.3)
  Cmax of 4-oxotretinoin | 3.14 (0.902) | 7.65 (0.732)

4. Secondary Outcome: A Summary of Pharmacokinetic Parameters (AUC0-t) After Single Dose of HF1K16
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | HF1K16-3mg/m² | HF1K16-6mg/m²
Number analyzed (Participants) | 6 | 6
h*ng/mL
  AUC(0-last ) of tretinoin | 469 (93.3) | 810 (113)
  AUC(0-last ) of 4-oxotretinoin | 2.58 (1.78) | 9.24 (3.21)

5. Secondary Outcome: A Summary of Pharmacokinetic Parameters (Tmax) After Single Dose of HF1K16
Description: o evaluate pharmacokinetic parameters of free tretinoin and liposome encapsulated tretinoin (4-oxotretinoin) in plasma after single administration of HF1K16
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: h
Arm/Group | HF1K16-3mg/m² | HF1K16-6mg/m²
Number analyzed (Participants) | 6 | 6
h
  Tmax of tretinoin | 0.92 [0.92 to 0.92] | 0.92 [0.92 to 0.93]
  Tmax of 4-oxotretinoin | 1.5 [1.5 to 2.0] | 1.8 [1.5 to 2.0]

ADVERSE EVENTS:
Time Frame: All AEs (serious and non-serious) were collected from signing the ICF and throughout the study to the follow-up/completion visit. A follow-up telephone call was placed to all subjects on Day 8 (± 2 days) to collect adverse event (AE) and concomitant medication information.
Groups:
- 3 mg/m² HF1K16: Cohort 1: enrolled 6 subjects for 3 mg/m2 of HF1K16
- 6 mg/m² HF1K16: Cohort 2: enrolled 6 subjects for 6mg/m2 of HF1K16
- Placebo: Cohort 1: enrolled 2 subjects for placebo Cohort 2: enrolled 2 subjects for placebo
Arm/Group | 3 mg/m² HF1K16 | 6 mg/m² HF1K16 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 4/6 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg/m² HF1K16 (N=6) | 6 mg/m² HF1K16 (N=6) | Placebo (N=4)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT05386823/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT05386823/SAP_001.pdf